CLINICAL TRIAL: NCT06844682
Title: The Effect of the Posıtıon Gıven to Patıents After Coronary Angıography on Back Paın and Comfort
Brief Title: Effect of Position on Back Pain and Comfort After Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Eyüp Fırat, Nurse, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AIBU-SBF-EF-01
Record Dates: First submitted 2024-11-14; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2024-11

CONDITIONS: Coronary Angiography

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Patients were assigned to the control and intervention groups by the minimization method. (Minimization was carried out according to parameters such as age, gender, and body mass index (BMI).
  A computer program that generates random numbers was used for the randomization process. In accordance with the randomization list, patients were randomly divided into intervention group and control group according to the order of admission to the hospital.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): At the end of CAG, the patients were laid in the supine position in line with the routine practice of the clinic and were allowed to remain in this position for 6 hours. While lying in bed, the patient identification form and VAS for comfort and pain were applied (Hour 0). VAS was applied at the 2nd and 4th hours following the removal of the mattresses. The patients' back pain and comfort were evaluated and the results were recorded on the relevant forms.
- intervention group (Experimental): After CAG, the patients were placed on the bed in the supine position. The first measurement was taken when he was put to bed after CAG, and the patient introduction form and VAS for comfort and pain were applied (0th hour). Following the removal of the mattresses, the patient was placed in the semi-fawler position. VAS was applied 2 and 4 hours after positioning. The patients' back pain and comfort were evaluated with the given position, and the results were recorded on the relevant forms.
  Interventions: Other: intervention group

INTERVENTIONS:
Other: intervention group — Following the removal of the mattresses, the patient was placed in the semi-fawler position.
  Arms: intervention group

SUMMARY:
After coronary angiography, back pain and comfort levels were measured while the intervention group was positioned and the control group was not positioned

DETAILED DESCRIPTION:
Patients were assigned to the control and intervention groups by the minimization method. Data were collected using the Visual Analog Scale (VAS) and a Patient Introduction Form to assess the pain and comfort levels of the patients. Prior to the starting the research, the necessary permissions were obtained from the institution where the study was conducted, from the patients and the ethics committee. In the analysis of data, frequency and percentage values, Kolmogorov-Smirnov test for the normal distribution of continuous variables, chi-square for comparisons of qualitative variables, two-way analysis of variance for comparison of repeated measurements of pain and comfort scores according to groups, and the relationship between two continuous variables were evaluated with the Pearson correlation coefficient. p<0.05 was considered statistically significant. IBM SPSS Statistics 23 package program was used for the analysis of the date. The intervention group was hospitalized in supine position after coronary angiography. The first measurement was taken when the patient was placed in bed after the procedure, and the Patient Introduction Form and VAS for comfort and pain were applied (Hour 0). Following the withdrawal of the mattresses, the patient was given the semi-fowler position. VAS was applied at the 2nd and 4th hours after the positioning. Patients in the control group were placed to bed in the supine position in accordance with the routine practice of the clinic at the exit of coronary angiography and were allowed to stay in this position for six hours. When the patients were put to in bed, the Patient Introduction Form, VAS were applied for comfort and pain (0. hour). VAS was applied at the 2nd and 4th hours following the removal of the mattresses. Patients' back pain and comfort were evaluated, and the results were recorded on the relevant forms.

ELIGIBILITY:
Inclusion Criteria:

* Coronary angiography for the first time in the coronary intensive care unit and cardiology clinic
* Volunteer to participate in the study
* Femoral angiography procedure performed
* It created patients who had no obstacle to communication.

Exclusion Criteria:

* More than one coronary angiography procedure was performed
* Not volunteering to participate in the study
* Radial angiography procedure was performed
* Having a history of back surgery, existing hernia, or chronic waist or back pain

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
control group | three months
  Patients were put to bed in the supine position at the exit of the CAG in accordance with the routine practice of the clinic and were allowed to stay in this position for 6 hours. When the patient was put to bed, VAS was applied for the patient introduction form, comfort and pain (0. hour). 2 From the withdrawal of mattresses. and 4. during the hours, VAS was applied. The patients' back pain and comfort were evaluated and the results were recorded in the relevant forms.
intervention group | three months
  The patients were put to bed after KAG. The first measurement was taken when he was put to bed after KAG. The patient introduction form, VAS were applied for comfort and pain (0. At sa Tu). Following the withdrawal of the mattresses, the patient was given the semi-fawler position. 2 After being given the position. and 4. hours later, VAS was applied. The back pain and comfort of the patients were evaluated with the given position and the results were recorded on the relevant forms.

CONTACTS AND LOCATIONS:
Overall Officials: Eyüp FIRAT, Principal Investigator — SANKO Üniversitesi
Locations (1):
- Eyüp, Gaziantep, şahinbey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No